CLINICAL TRIAL: NCT02019784
Title: A Placebo Controlled Single Centre Double Blind Randomised Trial to Investigate the Efficacy of Rifaximin Versus Placebo in Improving Systemic Inflammation and Neutrophil Malfunction in Patients With Cirrhosis and Chronic Hepatic Encephalopathy
Brief Title: Randomised Controlled Trial of Mechanistic Effects of Rifaximin in Cirrhosis and Chronic Hepatic Encephalopathy
Acronym: RIFSYS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: KCH14-183_RIFSYS_V4.0; 2013-004708-20 (EudraCT Number)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Liver Cirrhosis; Hepatoencephalopathy, Early Fatal Progressive
Keywords: Cirrhosis; Hepatic encephalopathy
MeSH Terms: conditions — Liver Cirrhosis; Combined Oxidative Phosphorylation Deficiency 1; Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin-α (Active Comparator): Rifaximin-α (TARGAXAN TM, manufactured by Alfa-Wasserman, Bologna, Italy) tablets - 550mg twice daily for 90 days
  Interventions: Drug: Rifaximin-α
- Placebo (Placebo Comparator): Placebo tablets - 550mg twice daily for 90 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Rifaximin-α — Rifaximin-α will be compared to placebo with the various outcome measures assessed at baseline (pre-randomisation), and then at 30 days and 90 days.
  Other Names: Targaxan (brand name)
  Arms: Rifaximin-α
Drug: Placebo Oral Tablet — Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
Patients with cirrhosis are particularly prone to infection which is frequently a precipitant of hepatic encephalopathy, renal failure and circulatory collapse. Bacterial infections are of particular concern in patients with cirrhosis because they are poorly tolerated. Sepsis and associated endotoxaemia whereby bacteria produce inflammatory particles occur in approximately 40% of hospitalized patients with cirrhosis and is a major cause of death.

Gut-derived and blood-borne pathogens can induce an inflammatory response within the liver and spleen, which are the major organs that remove bacteria and their endotoxin (such as lipopolysaccharide - LPS and bacterial DNA itself) from the bloodstream. Several mechanisms have been identified and proposed in this process which depends upon a balance between the barrier functions of the gut and the 'detoxifying' capacity of the liver. People with established liver cirrhosis have been shown to have escape of endotoxin into the bloodstream produced by bacteria that reside in their intestines, which becomes more permeable or 'leaky'.

Gut dysfunction is defined by changes in the types of bacteria within the gut and in overall permeability allowing bacterial products which would otherwise be contained within the gut to travel into the bloodstream and lymphatic system with detrimental effects elsewhere in the body. This passage of bacterial products is termed bacterial translocation, and it's effects on the liver and general immune system can be then be measured.

It has now become recognised that certain types of white blood cells such as neutrophils and monocytes become dysfunctional and this predisposes to infection and may also have a more direct pathogenic role in hepatic encephalopathy. Thus neutrophil and monocytes may be a novel pharmacotherapeutic target in a condition where current therapies such as bowel aperients (e.g. lactulose) are inadequate. A therapeutic strategy utilising Rifaximin, a non-absorbable antibiotic, to modulate gut bacterial which produce ammonia, a chemical known to be important in the cause of hepatic encephalopathy, could potentially lower gut-derived systemic inflammation, endotoxaemia, infection and organ dysfunction in this population improving outcomes and prolonging transplant-free survival.

We therefore plan to test if Rifaximin positively affects markers of immune dysfunction in patients with liver cirrhosis experiencing chronic hepatic encephalopathy after 30 days of treatment, as our primary research question.

Positive results from this study would support further trials into the potential benefit of using Rifaximin to improve immune function, as well as reduce the recurrence of hepatic encephalopathy, in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Overview

The study will be designed and conducted as a double blind placebo controlled randomised controlled trial - Clinical Trial of an Investigational Medicinal Product.

This study will be performed on patients referred to King's Liver Unit for further assessment and management of chronic overt hepatic encephalopathy (≥ Grade 1) or with ≥2 episodes of overt hepatic encephalopathy in the previous 6 months.

The study will be performed on 50 patients with cirrhosis and chronic hepatic encephalopathy [25 Rifaximin and 25 placebo] aged between 18 and 75 years managed within the Liver Unit at King's College Hospital which is the largest tertiary Liver Transplant Centre within the UK. For the purposes of this study a patient will be considered to have cirrhosis if they fulfil 2 out of 3 diagnostic criteria of confirmatory liver histology, biochemistry and/or radiologic findings consistent with cirrhosis/portal hypertension, and are presenting with chronic persistent overt hepatic encephalopathy (≥ grade 1) or with ≥2 episodes of overt hepatic encephalopathy in the previous 6 months.

Patient demographics, clinical details (including Westhaven hepatic encephalopathy grade) and blood haematology, biochemistry (including venous ammonia), microbiology data and neutrophil function will be assessed and collated at baseline and following 30 and 90 days of Rifaximin therapy or placebo. Intestinal permeability will be assessed using the intestinal disaccharide test. Faecal microbiota analysis will be performed by deep pyrosequencing techniques and plasma endotoxemia will be measured (lipopolysaccharide levels) with bacterial DNA quantification as a marker of bacterial translocation. These will all be measured at 3 time points: baseline and at 30 and 90 days after initiation of Rifaximin therapy or matching placebo.

Investigations

Patients will undergo intestinal functional tests within 7 days of recruitment, whereby they will be administered a test solution of not more than a cupful (150mls) of different types of non-absorbable sugars, which are drunk in liquid form by the participants. Prior to ingestion, baseline samples will be obtained as follows:

i) blood samples - for analysis of intestinal & immune (dys)function, and metabonomic analysis ii) urine sample - for intestinal (dys)function & metabonomic analysis iii) stool sample - for faecal biomarker and microbiota analysis

1v) ascitic sample (if clinically indicated) - surplus fluid will be analysed for bacterial translocation and immune (dys)function

Once the test solution has been ingested, blood samples will be obtained via a cannula which is placed in a vein, usually in the arm, prior to the start of the test, to allow further sampling without causing discomfort to the patient. A total of 15 samples will be obtained over a 5 hour period, with intervals ranging between 20-30mins, of not more than 6mls per sample. At the end of the test, at a 5 hour interval, a further urine sample will be collected to allow for intestinal functional testing. This is exactly the same procedure as that specified in the approved 'The Gut-Liver Axis in Liver Disease & Liver Transplantation' study (REC ref: 12/LO/1417).

Where participants are undergoing sampling of ascitic fluid for clinical reasons any fluid in excess of pathology's requirements will be analysed along with peripheral blood samples. Ascitic samples will only be taken from patients in whom a decision has been made to take these samples for clinical reasons (this decision will not be that of the investigator). No increased volume of such sample would be required.

Clinical outcomes (development of recurrent overt hepatic encephalopathy, organ failure and infection) will be recorded for a total of 90 days.

Analysis of samples - sites

Blood, urine and ascitic samples will be analysed in the Institute of Liver Studies and King's College Hospital laboratories where various tests to determine intestinal and immune function will be undertaken. Stool samples will be analysed both at laboratories at King's College Hospital and at the Franklin-Wilkins Building, King's College London, where faecal biomarkers and faecal microbiota analyses will be performed, respectively. Metabolic analyses for metabonomic profiling will be carried out at Imperial College London (both at St Mary's Hospital and at the South Kensington Campus).

Protocol

A more detailed list of the tests and analyses to be performed is to be found in the protocol. Study-specific flow charts have also been provided for a step-by-step representation of the study, visually representing the study process including participant recruitment, randomisation, sampling protocols and analyses at the three time points and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established cirrhosis complicated by hepatic encephalopathy
* For the purposes of this study a patient will be considered to have cirrhosis if they fulfil two out of the three diagnostic criteria of confirmatory liver histology, biochemistry and/or radiologic findings consistent with cirrhosis/portal hypertension, and
* are presenting with chronic persistent overt hepatic encephalopathy (≥ grade 1) or with ≥2 episodes of overt hepatic encephalopathy in the previous 6 months.

Exclusion Criteria:

* Age ≤18 or ≥75.
* Evidence of disseminated malignancy.
* Known coeliac or inflammatory bowel disease.
* Evidence of intestinal failure, intestinal obstruction and / or previous bowel resection.
* Pre-existing immunosuppressive states including HIV infection and chronic granulomatous diseases.
* Anti-inflammatory drug use e.g non-steroidals and immunomodulatory drug use e.g. prednisolone and azathioprine.
* Known hypersensitivity to rifaximin or rifamycin-derivatives
* Already receiving concomitant oral or parenteral antibiotic therapy e.g norfloxacin.
* Infection with clostridium difficile or stool testing positive for clostridium difficile toxin in the previous 3 months.
* Pregnancy or breast feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Rifaximin-α reducing neutrophil spontaneous oxidative burst ex vivo | Three time points: baseline before commencement of active drug/placebo, at 30 days and at 90 days
  To test whether there is a reduction in spontaneous neutrophil oxidative burst of 50% compared to baseline (as measured by the Burstest which measures the spontaneous production of reactive oxygen species) 30 days following the start of rifaximin-α/placebo therapy.

SECONDARY OUTCOMES:
Neutrophil bacteriocidal capacity | Three time points: baseline before commencement of active drug/placebo, at 30 days and at 90 days
  An improvement in neutrophil bacteriocidal capacity as measured by the Phagotest which utilises opsonised E. coli at 30 and 90 days
Reduction in systemic inflammation | Three time points: baseline before commencement of active drug/placebo, at 30 days and at 90 days
  A reduction in systemic inflammation as measured by plasma endotoxemia, bacterial DNA quantification and plasma pro-inflammatory cytokine profile at 90 days.
Improvement in neutrophil phenotype and function | Three time points: baseline before commencement of active drug/placebo, at 30 days and at 90 days
  An improvement in neutrophil phenotype and function including baseline and LPS-induced toll-like receptor 4 expression and intracellular cytokine production at 30 and 90 days.
Alterations in faecal microbiota at 90 days | Three time points: baseline before commencement of active drug/placebo, at 30 days and at 90 days
Reduction in intestinal permeability and changes in faecal biomarkers (calprotectin) at 90 days. | Three time points: baseline before commencement of active drug/placebo, at 30 days and at 90 days
Changes in urinary and plasma metabonomic profile | Three time points: baseline before commencement of active drug/placebo, at 30 days and at 90 days
  Changes in urinary and plasma metabonomic profile as measured by proton MR spectroscopy at 90 days

OTHER OUTCOMES:
Development of recurrent overt hepatic encephalopathy, organ failure and infection during the 90 day follow up | Three time points: baseline before commencement of active drug/placebo, at 30 days and at 90 days
Improvement in Trails A and B neuropsychiatric test score at 30 and 90 days. | Three time points: baseline before commencement of active drug/placebo, at 30 days and at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Shawcross, MBBS PhD, Principal Investigator — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, London, United Kingdom

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180
- [Derived] Patel VC, Lee S, McPhail MJW, Da Silva K, Guilly S, Zamalloa A, Witherden E, Stoy S, Manakkat Vijay GK, Pons N, Galleron N, Huang X, Gencer S, Coen M, Tranah TH, Wendon JA, Bruce KD, Le Chatelier E, Ehrlich SD, Edwards LA, Shoaie S, Shawcross DL. Rifaximin-alpha reduces gut-derived inflammation and mucin degradation in cirrhosis and encephalopathy: RIFSYS randomised controlled trial. J Hepatol. 2022 Feb;76(2):332-342. doi: 10.1016/j.jhep.2021.09.010. Epub 2021 Sep 24. PMID 34571050